CLINICAL TRIAL: NCT03146676
Title: The Ohio State University Dermatology Biorepository
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ben H Kaffenberger, Dermatologist, Ohio State University
Other Study IDs: 2010H0331
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin Tissue, Peripheral blood mononuclear cells, skin swabs, and saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will create and extend a source of clinical specimens for the future study of inflammatory skin disorders.

DETAILED DESCRIPTION:
A variety of molecular techniques can be used to investigate diseases by analyzing protein, DNA, and RNA. Flow cytometry, Polymerase chain reaction (PCR), histology and immunohistochemistry are assays which can identify specific cell populations and provide valuable information regarding the pathologic characteristics of those populations. Flow cytometry analyzes the surface markers of cells. Histology and immunohistochemistry further characterize surface and cellular molecules and aid in the diagnosis of certain skin diseases. Gene expression profiling allows investigators to examine the genes detectable to determine the function of the cells involved, and PCR techniques are useful for the diagnosis of certain conditions and for DNA analysis.

By procuring blood, skin tissue, and swab samples from patients with and without neoplastic and inflammatory skin disorders at the time of their appointments, the hypothesize that future translational research can be conducted on such specimens using the aforementioned techniques to further understand disease mechanisms in cutaneous disorders, and to potentially discover defective function and genetic mutations within cells from patients with neoplastic and inflammatory skin disorders. By establishing a tissue bank, we aim to lay the foundation for future work that will improve our understanding of the biology and natural history of neoplastic and inflammatory cutaneous diseases.

ELIGIBILITY:
Inclusion Criteria:

* Seen by an Ohio State University (OSU) Dermatology provider on the main University Hospital campus, including the James Cancer Hospital, OSU Dermatology East, OSU Dermatology at the Ohio State Eye and Ear Institute, Martha Morehouse Medical Pavilion, and OSU Dermatology at Upper Arlington after the date of approval of this protocol
* Ability to provide informed consent, or parent or legal guardian capable of providing consent for child or mentally handicapped individuals
* Willingness to participate in a research study.

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any person that meets the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Source of clinical specimens for the future study of neoplastic and inflammatory skin disorders | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kaffenberger, MD, Principal Investigator — Dermatologist
Locations (1):
- OSU Dermatology West, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No